CLINICAL TRIAL: NCT03729713
Title: Computerized Cognitive Rehabilitation in MS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Horizon Blue Cross Blue Shield of New Jersey (Other)
Responsible Party: Principal Investigator, Vikram Bhise, MD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018001642
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Computerized Cognitive Rehabilitation
  Interventions: Other: Computerized cognitive rehabilitation
- Placebo (Sham Comparator): Video game
  Interventions: Other: Sham placebo

INTERVENTIONS:
Other: Computerized cognitive rehabilitation — 6 week course of cognitive rehabilitation focused on attention, learning, and memory
  Arms: Intervention
Other: Sham placebo — an alternative home-based computer program not designed for cognitive remediation but of the same duration
  Arms: Placebo

SUMMARY:
This study examines a home-based computerized cognitive rehabilitation intervention in adults with multiple sclerosis compared to placebo (videogame). Patients are assessed through pre-and post neuropsychological testing.

DETAILED DESCRIPTION:
Patients will be randomized to enter a 6 week course of computer based cognitive rehabilitation focused on improving attention, learning, and memory. Control patients will receive an alternative home-based computer program not designed for cognitive remediation but of the same duration.

The primary outcome will be performance on neuropsychological testing in the intervention sample compared to controls. Secondary outcomes will be the measures of self-efficacy, work productivity, quality of life, fatigue, depression, anxiety, and healthcare utilization. Healthcare utilization variables include annual total cost (current year and prior), number and cost of ER/hospital/outpatient visits, number of hospital visits, hospital length of stay, number preventive visits, total number claims, and number of new medications initiated. In addition, acute changes in neuropsychological testing induced by a bout of physical activity (i.e. self-paced walking during the Six-Minute Walk Test) will be examined, and that pattern of change will be compared between intervention and control groups at each data collection point.

Each subject will participate for a total of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of multiple sclerosis with cognitive complaint

Exclusion Criteria:

1. Patients unwilling to participate
2. Patients who cannot attend NPT sessions
3. Patients with severe cognitive impairment
4. Non-English speaking patients (testing materials are in English)
5. Patients with intact neuropsychological functioning at baseline on testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive Functioning | 6 Months
  Compare between groups differences in attention (auditory and visual working memory), processing speed (automatic and controlled speed), executive functioning (verbal fluency and mental flexibility), and memory (immediate and delayed verbal and visual modalities) at completion of intervention, 3 months and 6 months using standardized scores.

SECONDARY OUTCOMES:
Multiple Sclerosis Self-Efficacy Scale | 6 Months
  Measures the person's perspective on maintenance and control over their multiple sclerosis
Work Productivity and Activity Impairment Instrument | 6 months
  Measures a person's impairments in their ability to work and participate in chosen activities
Multiple Sclerosis Quality of Life Inventory | 6 months
  A battery of quality of life scales designed for use by people with MS
Hospital Anxiety and Depression Scale | 6 months
  Measures depression and anxiety
Healthcare Utilization | 12 Months
  Compare between group differences in annual cost of care, ER visits, hospital visits, hospital length of stay, number of preventive visits, total number of claims, and neurology office visits

OTHER OUTCOMES:
Six-minute Walk Test | 6 months
  A measure of walking endurance - measures how far a person can walk in six minutes
Timed Up & Go Test | 6 months
  A timed test of functional mobility that tests a persons ability to stand, walk a short distance and return to sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No